CLINICAL TRIAL: NCT01967264
Title: A Randomized, Double Blind, Placebo Controlled Study to Evaluate the Safety Profile and Pharmacokinetic Parameters of Udenafil 150 mg in Healthy Mexican Subjects.
Brief Title: Safety and Pharmacokinetic Profile of Udenafil in Healthy Mexican Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: PK-MX031; U1111-1146-1315 (Other: World Health Organization)
Record Dates: First submitted 2013-10-17; First posted 2013-10-22 (Estimated); Last update posted 2013-10-22 (Estimated); Status verified 2013-10

CONDITIONS: Erectile Dysfunction; Phosphodiesterase 5 Inhibitor
Keywords: Drug therapy
MeSH Terms: conditions — Erectile Dysfunction | interventions — udenafil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Udenafil 150 mg + Udenafil 150 mg (Experimental): Udenafil 150 mg, tablet, orally, once on Day 1, followed by udenafil 150 mg, tablet, orally, once on Day 3.
  Interventions: Drug: Udenafil
- Udenafil 150 mg + Placebo (Experimental): Udenafil 150 mg, tablet, orally, once on Day 1, followed by placebo, tablet, orally, once on Day 3.
  Interventions: Drug: Udenafil; Drug: Placebo
- Placebo + Udenafil 150 mg (Experimental): Placebo, tablet, orally, once on Day 1, followed by udenafil 150 mg, tablet, orally, once on Day 3.
  Interventions: Drug: Udenafil; Drug: Placebo
- Placebo + Placebo (Placebo Comparator): Placebo, tablet, orally, once on Day 1, followed by placebo, tablet, orally, once on Day 3.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Udenafil — Udenafil tablets
  Arms: Placebo + Udenafil 150 mg; Udenafil 150 mg + Placebo; Udenafil 150 mg + Udenafil 150 mg
Drug: Placebo — Placebo tablets
  Arms: Placebo + Placebo; Placebo + Udenafil 150 mg; Udenafil 150 mg + Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of Udenafil 150 mg compared to placebo.

DETAILED DESCRIPTION:
The drug being tested in this study is called Udenafil. Udenafil is being tested to determine a safe and well-tolerated dose. This study will look at vital signs, laboratory tests and side effects in people who take Udenafil.

The study will enroll approximately 84 patients. Participants will be randomly assigned (by chance) and by blocks to assure balanced groups (i.e. same number of participants) to one of the four treatment schemes-which will remain undisclosed to the patient and study doctor during the study (unless there is an urgent medical need):

* a) Udenafil-Udenafil
* b) Udenafil- Placebo
* c) Placebo-Udenafil
* d) Placebo-Placebo

All participants will be asked to take one tablet on Day 1 and one tablet on Day 3.

This single-centre trial will be conducted in Mexico. The overall time to participate in this study is up to 7 days. Participants will make 3 visits to the clinic, including 5 days confinement to the clinic, and will be contacted by telephone 15 days after last visit to the clinic for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Sign a letter of informed consent prior to performing any procedure.
2. Male
3. Clinically healthy
4. Age between 18 and 55 years old.
5. Body Mass Index (BMI) between 18.5 and 24.9.
6. Capability and disposition to attend clinical intervention period

Exclusion Criteria:

1. Current use of any allopathic, over the counter (OTC) (e.g. nutritional supplements) or alternative (e.g. herbal) medication within two weeks prior to trial initiation.
2. History of psychiatric diseases.
3. History of drug abuse (alcohol, tobacco or any other).
4. Chronic consumption of caffeine (coffee, cola, green tea, St. Johns Wort).
5. Laboratory tests with clinically significant alterations.
6. Intestinal disorders that may modify absorption.
7. History of allergy to the drug or related drugs.
8. Blood donation within 45 days prior to study initiation.
9. Participation in a clinical trial within 2 months prior to study initiation.
10. History of orthostatic alterations or presyncope.
11. Vegetarian diet or other peculiar dietary habits which would interfere the participant's acceptance to standardized meals.
12. Inability to communicate or social vulnerability.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2013-07; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Participants with Adverse Events | 3 Weeks
  AEs will be evaluated by monitoring participants vital signs, laboratory tests (blood chemistry, hematology, coagulation and serology tests, urianalysis), electrocardiography (ECG).

SECONDARY OUTCOMES:
AUC(0-last): Area Under the Plasma Concentration-Time Curve From Time 0 to the Last Measured Concentration Above the Lower Limit of Quantification | Predose and at 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 5, 7, 9, 12, 24, 36 and 48 hours post-dose
  AUC(0-last) is a measure of total plasma exposure to the drug from Time 0 to the last measured concentration above the lower limit of quantification (LLOQ).
AUC(0-inf): Area Under the Plasma Concentration-time Curve from Time 0 to Infinity | Predose and at 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 5, 7, 9, 12, 24, 36 and 48 hours post-dose
  Area under the plasma concentration-time curve from time zero extrapolated to infinity.
Cmax: Maximum Observed Plasma Concentration | Predose and at 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 5, 7, 9, 12, 24, 36 and 48 hours post-dose
  Maximum observed plasma concentration (Cmax) is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve.
Tmax: Time to Reach the Maximum Plasma Concentration | Predose and at 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 5, 7, 9, 12, 24, 36 and 48 hours post-dose
  Time to reach the maximum plasma concentration (Cmax), equal to time (hours) to Cmax.
Terminal Phase Elimination Half-life (T1/2) | Predose and at 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 5, 7, 9, 12, 24, 36 and 48 hours post-dose
  Terminal phase elimination half-life (T1/2) is the time required for half of the drug to be eliminated from the plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (1):
- Querétaro, Mexico